CLINICAL TRIAL: NCT05661773
Title: Assessing the Effect of Vacuum Suction on Digital Ischemia in Critically Ill Patients
Brief Title: Digital Ischemia Reduction in Critically Ill Patients
Acronym: DIR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA required a new investigational device disclosure for using the wound vac in a new way
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00089927
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-06

CONDITIONS: Hypovolemic Shock; Cardiogenic Shock; Digital Ischemia
MeSH Terms: conditions — Shock; Shock, Cardiogenic

STUDY DESIGN:
Intervention Model Description: Each patient will act as their own control. By applying the vacuum assisted warmer to one hand, results can be compared to the contralateral hand. In this way, patient outcomes can be assessed between patients and indexed to each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- combined use of vacuum assisted suction and heat exchanger warming (Experimental): The novel idea that this study proposes, is the combined use of vacuum assisted suction and heat exchanger warming. It is well known that heat causes capillary vasodilation, where warming hands and toes improves blood flow while cooling them causes vasoconstriction. Applying a vacuum across a capillary bed increases the transcapillary gradient increasing the driving force of blood flow into tissues. The combination of these two mechanisms can work synchronously to improve blood flow to ischemic extremities and digits.
  Interventions: Device: the combined use of vacuum assisted suction and heat exchanger warming
- expectant medical management (No Intervention): expectant medical management will continue to the contralateral hand

INTERVENTIONS:
Device: the combined use of vacuum assisted suction and heat exchanger warming — Heat causes capillary vasodilation, where warming hands and toes improves blood flow while cooling them causes vasoconstriction. Applying a vacuum across a capillary bed increases the transcapillary gradient increasing the driving force of blood flow into tissues. The combination of these two mechanisms can work synchronously to improve blood flow to ischemic extremities and digits.
  Arms: combined use of vacuum assisted suction and heat exchanger warming

SUMMARY:
Patients requiring high dose pressors (minimum 2) who are unlikely to be weaned off them over 1 day will be identified. Patients will have the device applied to one hand while expectant medical management will continue to the contralateral hand.

DETAILED DESCRIPTION:
The proposed study offers no foreseeable risk to patients. The device relies on a wound vac system for vacuum generation which is industry standard and approved for creating safe suction applied to wounds. In this application, the same suction and device would be used to apply suction to an enclosure through which the hand is placed. Similarly, a heat exchanger would be used to run lukewarm water through a warming bad, which is technology that is routinely used in surgery. Heater coolers are used in every bypass surgery, and warming fluid blankets are common for helping to rewarm patients on the operating room table.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the cardiac critical care unit/cardiovascular intensive care unit with cardiac pathologies on vasopressor support

Exclusion Criteria:

* Patients who are not on vasopressor support
* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of digital ischemia | Day 14
  rate of digital ischemia characterized by tissue loss or destruction - measure incidence rate as a ratio of patients who got digital ischemia with the number of patients who were on vasopressors

SECONDARY OUTCOMES:
extent of digital ischemia - number of digits involved | Day 14
  extent of digital ischemia - determined by number of digits involved
extent of digital ischemia - length of digits involved | Day 14
  extent of digital ischemia - determined by degree of length of digits involved (like distal finger joint, proximal finger joint, entire finger, into the palm, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Bartlomiej Imielski, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No